CLINICAL TRIAL: NCT07110194
Title: Phase I Clinical Trial of TQB2825 Subcutaneous Injection in CD20-positive Hematological Malignancies
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Chia Tai Tianqing Pharmaceutical Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2825-I-02
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-05

CONDITIONS: CD20-positive Hematological Malignancies
MeSH Terms: interventions — Injections, Subcutaneous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2825 Injection (Subcutaneous Injection) (Experimental): The medication is administered once every two weeks, and the treatment lasts for 28 consecutive days, which constitutes one treatment cycle.
  Interventions: Drug: TQB2825 Injection (Subcutaneous Injection)

INTERVENTIONS:
Drug: TQB2825 Injection (Subcutaneous Injection) — TQB2825 is a Cluster of Differentiation 3 × Cluster of Differentiation 20 (CD3×CD20) dual antibody, which can simultaneously target the CD20 on tumor cells and the CD3 on T cells. It can induce T cell activation, proliferation and cytokine release, and effectively target and kill tumor cells.

SUMMARY:
The aim of this study is to evaluate the pharmacokinetic characteristics, safety and efficacy of the TQB2825 injection (subcutaneous administration) in patients with CD20-positive hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily participated in this study, signed the informed consent form, and had good compliance;
* Age 18 years or older and less than 80 years (calculated based on the date of signing the informed consent form);
* Eastern Cooperative Oncology Group (ECOG) score 0 to 2 points;
* Expected survival greater than 12 weeks;
* Malignant hematological tumors diagnosed by histological or cytological means, including diffuse large B-cell lymphoma, follicular lymphoma, mantle cell lymphoma, and marginal zone lymphoma, etc.;
* Immunophenotype analysis shows that the tumor is CD20 positive;
* Previously received at least one adequate treatment with a CD20 monoclonal antibody regimen (combined chemotherapy or single drug), and the most recent adequate treatment did not lead to remission or disease progression after remission, or relapsed after autologous hematopoietic stem cell transplantation (auto-HSCT);
* According to the 2014 Lugano criteria, there is at least one measurable lesion, that is, based on Computed Tomography (CT) cross-sectional images, the long diameter of lymph node lesions is greater than 15 mm or the long diameter of extranodal lesions is greater than 10 mm; Positron Emission Tomography - Computed Tomography scan (PET-CT) scan shows positive PET;
* Laboratory tests meet the following criteria (within 14 days before screening, no blood transfusion, no use of hematopoietic stimulating factors and other drugs to correct):

  1. Hemoglobin (HGB) ≥ 80 g/L;
  2. Absolute neutrophil count (NEUT) ≥ 1.0 × 109/L;
  3. Platelet count (PLT) ≥ 75 × 109/L (if accompanied by bone marrow invasion, platelet ≥ 50 × 109/L).
  4. Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN);
  5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 ULN. If accompanied by liver metastasis, then ALT and AST ≤ 5 ULN;
  6. Serum creatinine (CR) ≤ 1.5 ULN or estimated glomerular filtration rate by Cockcroft-Gault formula ≥ 50 ml/min.
  7. Prothrombin time (PT), activated partial thromboplastin time (APTT), and international normalized ratio (INR) ≤ 1.5 × ULN (not receiving anticoagulant treatment);
* Pregnant women should agree to use effective contraceptive measures during the study period and within 12 months after the study ends. For men, they should agree to use effective contraceptive measures during the study period and within 12 months after the study ends.

Exclusion Criteria:

* Within the 5 years prior to the first medication administration, the subject had or currently has other malignant tumors. The following two situations can be included in the study: other malignant tumors treated by a single surgical procedure, achieving 5 consecutive years of disease-free survival (DFS); cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumors), Tis (in situ cancer), and T1 (tumor infiltration of the basement membrane)];
* Previous treatment-induced adverse reactions have not recovered to a Common Terminology Criteria for Adverse Events, Version 5 (CTCAEv5.0) score of ≤1, except for grade 2 alopecia, non-clinically significant and asymptomatic laboratory abnormalities, stable thyroid function hypofunction after hormone replacement therapy, etc., which are judged by the investigator to have no safety risks;
* Previous anti-tumor treatment:

  1. Within 4 weeks before the first administration, received chemotherapy, immunotherapy, monoclonal antibody treatment, radiation therapy within 2 weeks, or small molecule targeted drugs, or still within the 5 half-lives of the drug (based on the earliest occurrence time), calculate the washout period from the end of the last treatment;
  2. Treatment with Chinese patent medicines (including Compound Banmao Capsules, Kang'ai Injection, Kanglaite Capsules/Injection, Aidi Injection, Yadanzi Oil Injection/Capsules, Xiaoaiping Tablets/Injection, Huachansu Capsules, etc.) that are explicitly approved by the National Medical Products Administration (NMPA) with anti-tumor indications in the package insert within 2 weeks prior to the first dose;
  3. Previously used other antibodies targeting both CD3 and CD20 for treatment;
  4. Received Chimeric Antigen Receptor T-cell (CAR-T) treatment, or other immune cell therapy, or autologous hematopoietic stem cell transplantation (auto-HSCT) within 3 months before the first administration;
* Lymphoma has previously or currently involved or is suspected to involve the central nervous system or lymphoma leukemia;
* Within 4 weeks before the first administration, received major surgical treatment, significant traumatic injury, or expected to undergo major surgery during the study treatment, or has long-standing unhealed wounds or fractures;
* Within 4 weeks before the first administration, experienced any bleeding or bleeding event ≥ Common Terminology Criteria for Adverse Events (CTC AE) 3 grade in the subject.
* Within 6 months before the first administration, had a thromboembolic event such as cerebral vascular accident (including transient ischemic attack), deep vein thrombosis, and pulmonary embolism, or any history of severe thromboembolism (implantable venous infusion port or catheter-related thrombosis, or superficial venous thrombosis is not considered "serious" thromboembolism);
* Has clinically significant uncontrolled need for repeated drainage of pleural effusion, ascites, or moderate or above pericardial effusion; Decompensated liver cirrhosis (Child-Pugh liver function rating of B or C) and active hepatitis (B).
* Pulmonary diseases, including any of the following conditions:

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Peak time | Up to 4 month
  Time to peak blood concentration after a single dose
Peak concentration Cmax | Up to 4 month
  After a single dose, the highest point of the drug-time curve is called the peak concentration.
Plasma elimination half-life t1/2 | Up to 4 month
  The amount of time it takes for the concentration of the drug in the blood, or the amount of drug in the body, to drop to about half of its original level.

SECONDARY OUTCOMES:
Incidence and severity of AE and Serious Adverse Event (SAE), and abnormal laboratory test indicators | Up to 24 month
  Incidence and severity of AE and SAE, and abnormal laboratory test indicators
Overall response rate | Up to 24 month
  To assess the percentage of patients with complete (CR) or partial response (PR) in the CD20-positive hematological tumor population who received the TQB2825 subcutaneous injection.
Complete response rate | Up to 24 month
  To evaluate the percentage of complete response (CR) achieved by the subcutaneous injection of TQB2825 in patients with CD20-positive hematological malignancies.
Progression-free survival period | Up to 24 month
  To evaluate the progression-free survival of TQB2825 subcutaneous injection in patients with CD20-positive hematological malignancies.
Duration of relief | Up to 4 month
  To evaluate the duration of remission of the TQB2825 subcutaneous injection in patients with CD20-positive hematological malignancies.
Overall survival period | Up to 4 month
  Evaluate the overall survival period of TQB2825 subcutaneous injection in patients with CD20-positive hematological malignancies.
Immunogenicity | Up to 8 month
  Evaluation of the immunogenicity data of TQB2825 subcutaneous injection in patients with CD20-positive hematological malignancies.
Receptor occupancy rate | Up to 6 month
  Evaluate the receptor occupancy rate of TQB2825 subcutaneous injection in patients with CD20-positive hematological malignancies.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China